CLINICAL TRIAL: NCT02761681
Title: Mindfulness and Acceptance Applied in Colleges Through Web-Based Guided Self-Help
Brief Title: Mindfulness and Acceptance Applied in Colleges Through Web-Based Guided Self-Help (Phase II)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Contextual Change LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R44AT006952 (NIH)
Record Dates: First submitted 2015-04-30; First posted 2016-05-04 (Estimated); Last update posted 2019-07-29 (Actual); Status verified 2019-07

CONDITIONS: Mental Health
Keywords: Acceptance and Commitment Therapy; Mindfulness; Guided self-help; College students; Focused Interviews; RCT Control Condition; RCT ACT-CL Condition
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ACT-CL Web-based guided self-help (Experimental): Behavioral: Experimental Web-based guided self-help Program This intervention will involve counselor training and student use of the developed program. Counselors will complete training and invite students to participate, and will monitor and guide students in completing the series of 8 web-based sessions based on Acceptance and Commitment Therapy.
  Interventions: Behavioral: ACT-CL Web-based guided self-help
- Control Web-based guided self-help (Active Comparator): Behavioral: Control Web-based guided self-help program This intervention will be created for the current study. It will involve psycho-education on how students might get the most out of counseling. Counselors will go through the psycho-education session before inviting students to participate.
  Interventions: Behavioral: Control Web-based guided self-help

INTERVENTIONS:
Behavioral: ACT-CL Web-based guided self-help
  Arms: ACT-CL Web-based guided self-help
Behavioral: Control Web-based guided self-help
  Arms: Control Web-based guided self-help

SUMMARY:
This study will develop and then test a web-based guided self-help version of Acceptance and Commitment Therapy (ACT) to be utilized at college counseling centers (CCCs). ACT is an evidence-based transdiagnostic therapy found to effectively treat a range of psychological problems. An ACT program would provide a means of implementing effective treatment for the range of problems in the CCC setting, while the guided self-help format would reduce counselors' workload, improving cost-effectiveness and reducing waiting lists. This would both treat students and train counselors in how to implement the ACT intervention.

DETAILED DESCRIPTION:
Nearly half of all college students have a diagnosable mental health problem. College counseling centers (CCCs) are faced with increasing demands for services from Universities, students, and parents to meet the treatment needs of their students, in the context of increasingly severe cases and declining resources. Innovative, cost effective solutions are needed that can improve treatment effectiveness with a range of presenting problems while reducing counselor workloads.

The current project seeks to meet these needs by building a user-informed guided self-help version of Acceptance and Commitment Therapy (ACT), an evidence-based transdiagnostic therapy that has been found to effectively treat a range of mental health problems by targeting experiential avoidance, the tendency to avoid unwanted emotions and negative thoughts.After the program has been built in the first stage of the study, the investigators will then test this program at several CCCs throughout the country. An ACT program would provide a means of implementing effective treatment for the range of problems encountered in the CCC setting, while the online guided self-help format would reduce counselors' workload for each client, improving cost effectiveness and reducing waiting lists. This product would both treat students through a series of self-help modules and train CCC counselors in how to implement the guided self-help ACT intervention.

For the current phase (Phase II) of this Small Business Innovation Research (SBIR) grant, 8 student self-help sessions will be developed, as well as a counselor portal with counselor training sessions to review students' use of the program and to receive training on implementing ACT guided self-help.

The current study will consist of two stages: Stage 1 will study user preferences and testing of the program as it is developed, and Stage 2 will be a randomized trial of the program in several CCCs.

Stage 1 will consist of ongoing interviews with a total of 6 students, 7 counselors and 1 director, who will be contacted intermittently throughout the program to participate in web-conference interviews in which they provide feedback on the current development, and test individual components of the program. Development will be iterative, and will be updated and adjusted based on the feedback from these focused interviews.

Stage 2 will consist of a randomized trial of 40 counselors using the program, and a nested program evaluation of 400 students (10 students per counselor). Counselors will be randomized to either the ACT on College Life program, or to a control website. After completing the condition's training, counselors will invite students to participate in the site to which the counselor has been randomized. Participants in both conditions will complete assessments at baseline, post, and follow-up. The study will examine the feasibility, efficacy, and acceptability of the program with both students and counselors.

ELIGIBILITY:
Inclusion Criteria:

* (Stage 1a: Counselor Focused Interviews): Currently working at CCC or previously worked at CCC for more than 1 year
* (Stage 1a: Counselor Focused Interviews): Willing to spend approximately 9 hours across 5-7 phone or web conferences discussing elements and content of the web-based program as modules are developed
* (Stage 1a: Counselor Focused Interviews): Participation will comply with targeted enrollment plans
* (Stage 1b: Student Focused Interviews): Currently being treated at a local CCC, and seen by a counselor for a minimum of 4 sessions.
* (Stage 1b: Student Focused Interviews): Between the ages of 18-25
* (Stage 1b: Student Focused Interviews): Willing to spend approximately 10 hours across 8-12 phone or web conference sessions discussing elements of content of the web-based, guided self-help program as modules are developed.
* (Stage 1b: Student Focused Interviews): Student is currently not suicidal or homicidal, and does not have a history of psychosis
* (Stage 1b: Student Focused Interviews): Participation will comply with targeted enrollment plans, which also include adequate representation of participants across various clinical presentations
* (Stage 1c: Director Focused Interviews): Currently working at a CCC as a director, or previously worked at a CCC as a director for more than 1 year
* (Stage 1b: Student Focused Interviews): Willing to spend approximately 9 hours across 5-7 phone or web conference sessions discussing elements and content of the web-based, guided self help program as modules are developed.
* (Stage 1b: Student Focused Interviews): Participation will comply with targeted enrollment plans.
* (Stage 2a: Counselor RCT): Currently working at a CCC that received internal/local IRB approval for this study
* (Stage 2a: Counselor RCT): Willingness to be randomized to either ACT+TAU or a Psychoeducation+TAU condition
* (Stage 2a: Counselor RCT): If randomized to ACT+TAU, willingness to take the ACT guided self-help training during the 4 weeks prior to the start of the Fall 2016 semester, until reaching a passing criterion of 80% (which will take approximately 9 hours)
* (Stage 2a: Counselor RCT): Willingness to attempt to recruit 10 student clients to participate either in the ACT self-help modules (if counselor is in ACT+TAU condition) or in the psychoeducation website (if counselor is in Psychoeducation+TAU)
* (Stage 2a: Counselor RCT): Willingness to monitor all student participants they recruit as long as students remain active participants (with the potential to de-activate students whose continued participation in the study may be contraindicated).
* (Stage 2a: Counselor RCT): Participation will comply with targeted enrollment plans
* (Stage 2b: Student Program Evaluation): Currently being treated at a CCC
* (Stage 2b: Student Program Evaluation): Students receiving counseling from ACT+TAU counselors: As covered on the consent form, willingness to participate in eight 30-minute modules as part of a web-based guided self-help program and complete pre- and post-assessments across a period of 10 weeks, OR Students receiving counseling from Psychoeducation+TAU counselors: As covered on the consent form, willingness to access psychoeducational website and complete three sets of questionnaires: one at the start of the study, another set 10 weeks later, and a follow-up set to 2 months after the post.
* (Stage 2b: Student Program Evaluation): Referred to study by counselor; cannot self-refer
* (Stage 2b: Student Program Evaluation): Student is clinically stable as per counselor judgment (e.g., not suicidal, psychotic, disruptive)
* (Stage 2b: Student Program Evaluation): Participation will comply with the targeted enrollment plans

Exclusion Criteria:

* (Stage 1a: Counselor Focused Interviews): Very uncomfortable with technology (Scoring 0-1 on a 0-5 Likert-like scale on comfort with web-based presentations)
* (Stage 1b: Student Focused Interviews): Under 18 years old
* (Stage 1b: Student Focused Interviews): Lack of fluency in English at the 7th grade level
* (Stage 1c: Director Focused Interviews): Very uncomfortable with technology (Scoring 0-1 on a 0-5 Likert-like scale on comfort with web-based presentations)
* (Stage 2a: Counselor RCT): None
* (Stage 2b: Student Program Evaluation): Under 18 years old
* (Stage 2b: Student Program Evaluation): Lack of fluency in English at the 7th grade level.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Change in Mental Health Symptoms - Counseling Center Assessment of Psychological Symptoms-62 | Baseline (week 1), Post (week 8), Follow-up (week 16)
  (Student Data) We will assess the change in various diagnoses and presentations common in college students (such as depression, anxiety, eating disorders, substance abuse, etc). This will be our primary outcome measure for students.

SECONDARY OUTCOMES:
System Usability Scale | Post (week 8 or week 20)
  (Counselor and Student Data) Program usability/acceptability will be a primary outcome
ACT Knowledge Questionnaire | Baseline (week 1) and post (week 20)
  (Counselor Data) We will examine whether counselors improve in their knowledge of ACT concepts after going through the program to assess initial feasibility of the prototype program.
Counselor Implementation Questions | Post (week 20)
  (Counselor Data) We will examine whether counselors were satisfied with the program utility, efficiency, and content and will explore the potential for subsequent dissemination of the website.
Personal Values Questionnaire | Baseline (week 1), Post (week 8) and Follow-up (week 16)
  We will examine whether students improve in their connection to and engagement in personal values after completing the program as a secondary process measure.
Satisfaction with Life Scale | Baseline (week 1), Post (week 8) and Follow-up (week 16)
  We will examine whether students improve on a measure of satisfaction with life after completing the program as a secondary outcome measure.
Acceptance and Action Questionnaire - II | Baseline (week 1), Post (week 8) and Follow-up (week 16)
  We will examine whether students improve on a measure of psychological flexibility after completing the program as a secondary process measure
Five Facet Mindfulness Questionnaire | Baseline (week 1), Post (week 8) and Follow-up (week 16)
  We will examine whether students improve on mindfulness variables (observing, acting with awareness, and being nonjudgmental) after using the program as a secondary process measure.
Acceptance and Action Questionnaire for University Students | baseline (week 1), post (week 8), follow-up (week 16)
  We will examine whether students improve on a measure of psychological flexibility tailored specifically to challenges college students experience as a secondary process measure
Satisfaction with Social Roles and Activities - Short Form Questionnaire | Baseline (week 1), Post (week 8) and Follow-up (week 16)
  PROMIS measure relating to satisfaction with participating in social roles and activities
Counseling Questions | Post (Week 8), and Follow-up (week 16)
  (Student Data) We will examine aspects of how the program was used in conjunction with counseling
Student Implementation and Satisfaction Questions | post (week 8) and follow-up (week 16)
  (Student Data) Assesses the user's satisfaction with and use of the program in the student counseling center context

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Pistorello, Principal Investigator — Contextual Change LLC; Michael Levin, Principal Investigator — Contextual Change LLC; Crissa Levin, Principal Investigator — Contextual Change LLC
Locations (1):
- Contextual Change, LLC, Reno, Nevada, United States

IPD SHARING:
Plan to Share IPD: No